CLINICAL TRIAL: NCT01258803
Title: A Randomized, Evaluator-Blind, Crossover, Single Dose Study of the Bronchodilator Effect of Formoterol Fumarate in Combination With Mometasone Furoate Metered Dose Inhaler Delivered With and Without a Spacer Versus Placebo and Foradil® Aerolizer® in Children With Persistent Asthma (Protocol No. P06476)
Brief Title: A Study of the Bronchodilator Effect of Formoterol Fumarate Used in Combination With Mometasone Furoate Metered Dose Inhaler in Children With Persistent Asthma (P06476 AM2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P06476; MK-0887A-178 (Other: Merck Research Laboratories)
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Asthma
Keywords: asthma; children; persistent
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): Treatment Period 1: Placebo MDI with spacer; Treatment Period 2: MF/F MDI without spacer; Treatment Period 3: MF/F MDI with spacer; Treatment Period 4: F DPI
  Interventions: Drug: Formoterol Fumarate DPI; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) without spacer; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) with spacer; Drug: Placebo MDI with spacer; Drug: Mometasone Furoate DPI
- Sequence 2 (Experimental): Treatment Period 1: F DPI; Treatment Period 2: MF/F MDI without spacer; Treatment Period 3: MF/F MDI with spacer; Treatment Period 4: Placebo MDI with spacer
  Interventions: Drug: Formoterol Fumarate DPI; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) without spacer; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) with spacer; Drug: Placebo MDI with spacer; Drug: Mometasone Furoate DPI
- Sequence 3 (Experimental): Treatment Period 1: MF/F MDI without spacer; Treatment Period 2: F DPI; Treatment Period 3: Placebo MDI with spacer; Treatment Period 4: MF/F MDI with spacer
  Interventions: Drug: Formoterol Fumarate DPI; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) without spacer; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) with spacer; Drug: Placebo MDI with spacer; Drug: Mometasone Furoate DPI
- Sequence 4 (Experimental): Treatment Period 1: Placebo MDI without spacer; Treatment Period 2: MF/F MDI with spacer; Treatment Period 3: F DPI; Treatment Period 4: MF/F MDI without spacer
  Interventions: Drug: Formoterol Fumarate DPI; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) without spacer; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) with spacer; Drug: Placebo MDI without spacer; Drug: Mometasone Furoate DPI
- Sequence 5 (Experimental): Treatment Period 1: MF/F MDI without spacer; Treatment Period 2: F DPI; Treatment Period 3: MF/F MDI with spacer; Treatment Period 4: Placebo MDI without spacer
  Interventions: Drug: Formoterol Fumarate DPI; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) without spacer; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) with spacer; Drug: Placebo MDI without spacer; Drug: Mometasone Furoate DPI
- Sequence 6 (Experimental): Treatment Period 1: MF/F MDI with spacer; Treatment Period 2: Placebo MDI without spacer; Treatment Period 3: MF/F MDI without spacer; Treatment Period 4: F DPI
  Interventions: Drug: Formoterol Fumarate DPI; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) without spacer; Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) with spacer; Drug: Placebo MDI without spacer; Drug: Mometasone Furoate DPI

INTERVENTIONS:
Drug: Formoterol Fumarate DPI — Two inhalations of Formoterol Fumarate DPI 10 mcg administered as a single dose
  Other Names: SCH 045571; MK-5571; Foradil® Aerolizer®
Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) without spacer — Two inhalations of Mometasone Furoate/Formoterol Fumarate MDI 50/5 mcg administered as a single dose without an AeroChamber Plus® Flow-Vu® Anti-Static Valved Holding Chamber (spacer)
  Other Names: SCH 418131; MK-0877A
Drug: Mometasone Furoate/Formoterol Fumarate MDI (ex-actuator) with spacer — Two inhalations of Mometasone Furoate/Formoterol Fumarate MDI 50/5 mcg administered as a single dose with an AeroChamber Plus® Flow-Vu® Anti-Static Valved Holding Chamber (spacer)
  Other Names: SCH 418131; MK-0877A
Drug: Placebo MDI with spacer — Two inhalations of placebo MDI administered as a single dose with an AeroChamber Plus® Flow-Vu® Anti-Static Valved Holding Chamber (spacer)
  Arms: Sequence 1; Sequence 2; Sequence 3
Drug: Placebo MDI without spacer — Two inhalations of placebo MDI administered as a single dose without an AeroChamber Plus® Flow-Vu® Anti-Static Valved Holding Chamber (spacer)
  Arms: Sequence 4; Sequence 5; Sequence 6
Drug: Mometasone Furoate DPI — Two inhalations of MF DPI 100 mcg administered as a single dose once daily at night. Used as maintenance therapy during screening and in between single doses of study drug.
  Other Names: SCH 032088; MK-0887; Asmanex® Twisthaler®

SUMMARY:
A study to compare the bronchodilatory effect of a single dose of Mometasone Furoate/Formoterol Fumarate (MF/F) pressurized metered dose inhaler (MDI) delivered with and without an AeroChamber Plus® with Flow-Vu® Anti-Static Valved Holding Chamber (spacer) versus Placebo MDI (combined with and without spacer) and formoterol fumarate (F) dry powder inhaler (DPI). Participants were randomly assigned to 1 of 6 treatment sequences and each participant was to receive a single dose of each of 4 treatments in each period. Each treatment period was separated by a 5 to 7 day washout period. It assumed that a single dose MF/F MDI 100/10 microgram (mcg) delivered with a spacer would produce bronchodilation, defined as a significant increase in forced expiratory volume in one second (FEV1) area under the curve from 0 to 12 hours (AUC[0-12 hr]) when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of asthma of at least 6 months duration
* Must have taken an Inhaled Corticosteroid ([ICS]; alone or in combination with a long-acting beta-2 Agonist [LABA]) for at least 3 months prior to the Screening Visit and must have been on a stable daily dose for at least 2 weeks prior to the Screening Visit
* FEV1 must be at least 70% predicted after all restricted medications have been withheld for the appropriate intervals
* Must demonstrate an increase in absolute FEV1 of at least 12% within 30 minutes after administration of 360 mcg albuterol (4 inhalations x 90 mcg, ex-actuator) or of nebulized albuterol (2.5 mg), if confirmed as standard office practice

Exclusion Criteria:

* Has been treated in the emergency room for a severe asthma exacerbation requiring systemic glucocorticosteroid treatment, or hospitalized for management of airway obstruction within 3 months prior to the Screening Visit
* Has required ventilator support for respiratory failure secondary to asthma
* Demonstrates a decrease in absolute FEV1 of >20% at any time from the Screening Visit up to and including the Baseline Visit
* Requires the use of greater than 8 inhalations per day of short-acting beta-2 agonists (SABA) MDI, or 2 or more nebulized treatments per day of 2.5 mg SABA on any 2 consecutive days from the Screening Visit up to and including the Baseline Visit
* Experiences a clinical deterioration in asthma that results in emergency treatment, hospitalization due to asthma, or treatment with additional, excluded asthma medication (including oral or other systemic corticosteroids, but allowing SABA) as judged by the investigator, at any time from the Screening Visit up to and including the Baseline Visit

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Teper, MD, Study Chair — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berger WE, Bensch GW, Weinstein SF, Skoner DP, Prenner BM, Shekar T, Nolte H, Teper AA. Bronchodilation with mometasone furoate/formoterol fumarate administered by metered-dose inhaler with and without a spacer in children with persistent asthma. Pediatr Pulmonol. 2014 May;49(5):441-50. doi: 10.1002/ppul.22850. Epub 2013 Sep 9. PMID 24019197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 28 study sites in the United States. Primary Therapy Period: December 2010 to October 2011.
Pre-assignment Details: The study included a 4-week Run-In Period during which participants were treated with Mometasone Furoate (MF) Dry Powdered Inhaler (DPI) 100 mcg.
Groups:
- Treatment Sequence 1: Treatment Period 1: Placebo Metered Dose Inhaler (MDI) with spacer, Treatment Period 2: Mometasone Furoate/Formoterol Fumarate (MF/F) MDI without spacer, Treatment Period 3: MF/F MDI with spacer, Treatment Period 4: F Dry Powder Inhaler (DPI)
- Treatment Sequence 2: Treatment Period 1: F DPI, Treatment Period 2: MF/F MDI without spacer, Treatment Period 3: MF/F MDI with spacer, Treatment Period 4: Placebo MDI with spacer
- Treatment Sequence 3: Treatment Period 1: MF/F MDI without spacer, Treatment Period 2: F DPI, Treatment Period 3: Placebo MDI with spacer, Treatment Period 4: MF/F MDI with spacer
- Treatment Sequence 4: Treatment Period 1: Placebo MDI without spacer, Treatment Period 2: MF/F MDI with spacer, Treatment Period 3: F DPI, Treatment Period 4: MF/F MDI without spacer
- Treatment Sequence 5: Treatment Period 1: MF/F MDI without spacer, Treatment Period 2: F DPI, Treatment Period 3: MF/F MDI with spacer, Treatment Period 4: Placebo MDI without spacer
- Treatment Sequence 6: Treatment Period 1: MF/F MDI with spacer, Treatment Period 2: Placebo MDI without spacer, Treatment Period 3: MF/F MDI without spacer, Treatment Period 4: F DPI
Period: Treatment Period 1 (1 Dose)
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started | 15 | 16 | 15 | 15 | 15 | 16
Completed | 15 | 16 | 15 | 15 | 15 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (1 Dose)
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started | 15 | 16 | 15 | 15 | 15 | 16
Completed | 14 | 14 | 15 | 15 | 15 | 15
Not Completed | 1 | 2 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (1 Dose)
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started | 14 | 14 | 15 | 15 | 15 | 15
Completed | 14 | 14 | 14 | 15 | 15 | 15
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 4 (1 Dose)
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started | 14 | 14 | 14 | 15 | 15 | 15
Completed | 14 | 14 | 14 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 92
Age, Customized [Number; unit: participants]
  5-7 years | 17
  8-11 years | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From 0-12 Hours (AUC[0-12h]) of the Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) After a Single Dose of MF/F MDI With Spacer Compared to Placebo MDI Combined With or Without Spacer
Description: The AUC was standardized to liters by dividing the length of time for which measurements of FEV1 were included in the calculation of the AUC. Baseline was defined as the average of 2 pre-dose FEV1 measurements (taken 30 minutes before and immediately before dosing), which was subtracted from each of the serial FEV1 measurements over the 12-hour period. The AUC was calculated based on these changes from the baseline evaluations using the trapezoidal rule.
Time Frame: Up to 12 hours postdose
Population: Participants who received each assigned single-dose treatment, performed at least the 0- and 2-hour spirometry evaluations and met the following criteria: did not use any prohibited concomitant medications; demonstrated satisfactory use of inhaler, spacer and spirometry maneuvers; and used >80% of prescribed MF DPI across the entire study treatment
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- MF/F MDI With Spacer: Participants receiving a single dose of MF/F MDI 100/10 mcg with a spacer
- Placebo MDI With or Without Spacer: Participants receiving a single dose of Placebo MDI with or without a spacer
Arm/Group | MF/F MDI With Spacer | Placebo MDI With or Without Spacer
Number analyzed (Participants) | 79 | 79
Liters | 0.115 (0.016) | -0.009 (0.016)
Statistical Analysis 1: Comparison: MF/F MDI With Spacer vs Placebo MDI With or Without Spacer; Pairwise Treatment Comparison of MF/F MDI with spacer and Placebo MDI combined with or without spacer. Analysis was performed using an analysis of covariance (ANCOVA) model extracting the effects due to treatment, sequence, subject (random effect nested within sequence), period, age groups (5 to 7 years and 8 to 11 years) and Baseline FEV1 as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.124, 95% CI 2-sided [0.094 to 0.154]

2. Secondary Outcome: AUC(0-12h) of the Change From Baseline in FEV1 After a Single Dose MF/F MDI Without Spacer Compared to Placebo MDI Combined With or Without Spacer
Description: as for outcome 1
Time Frame: Up to 12 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- MF/F MDI Without Spacer: Participants receiving a single dose of MF/F MDI 100/10 mcg without a spacer
Arm/Group | MF/F MDI Without Spacer | Placebo MDI With or Without Spacer
Number analyzed (Participants) | 79 | 79
Liters | 0.093 (0.016) | -0.009 (0.016)
Statistical Analysis 1: Comparison: MF/F MDI Without Spacer vs Placebo MDI With or Without Spacer; Pairwise Treatment Comparison of MF/F MDI without spacer and Placebo MDI combined with or without spacer. Analysis was performed using an ANCOVA model extracting the effects due to treatment, sequence, subject (random effect nested within sequence), period, age groups (5 to 7 years and 8 to 11 years) and Baseline FEV1 as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [0.073 to 0.131]

3. Secondary Outcome: AUC(0-12h) of the Change From Baseline in FEV1 After a Single Dose of MF/F MDI With Spacer Compared to MF/F MDI Without Spacer
Description: as for outcome 1
Time Frame: Up to 12 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | MF/F MDI With Spacer | MF/F MDI Without Spacer
Number analyzed (Participants) | 79 | 79
Liters | 0.115 (0.016) | 0.093 (0.016)
Statistical Analysis 1: Comparison: MF/F MDI With Spacer vs MF/F MDI Without Spacer; Pairwise Treatment Comparison of MF/F MDI with spacer and MF/F MDI without spacer. Analysis was performed using an ANCOVA model extracting the effects due to treatment, sequence, subject (random effect nested within sequence), period, age groups (5 to 7 years and 8 to 11 years) and Baseline FEV1 as a covariate; Test type: Superiority or Other; p = 0.144, ANCOVA; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.008 to 0.052]

4. Secondary Outcome: Change From Baseline in FEV1 After a Single Dose of MF/F MDI With Spacer, MF/F MDI Without Spacer, F DPI or Placebo MDI Combined With or Without Spacer at 5 and 30 Minutes, 1, 2, 4, 8 and 12 Hours Postdose
Description: Baseline was defined as the average of 2 predose measurements (taken 30 minutes and immediately before dosing).
Time Frame: Baseline and 5 and 30 minutes, 1, 2, 4, 8 and 12 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- F DPI: Participants receiving a single dose of F DPI 20 mcg
Arm/Group | MF/F MDI With Spacer | MF/F MDI Without Spacer | F DPI | Placebo MDI With or Without Spacer
Number analyzed (Participants) | 79 | 79 | 79 | 79
Liters
  Baseline (n=79, 79, 79, 79) | 1.554 (0.049) | 1.563 (0.049) | 1.570 (0.049) | 1.547 (0.049)
  5 minutes postdose (n=79, 79, 79, 79) | 0.111 (0.014) | 0.068 (0.013) | 0.105 (0.013) | -0.001 (0.014)
  30 minutes postdose (n=79, 79, 79, 79) | 0.131 (0.017) | 0.099 (0.016) | 0.117 (0.016) | 0.006 (0.016)
  1 hour postdose (n=79, 79, 79, 79) | 0.159 (0.017) | 0.131 (0.016) | 0.136 (0.016) | 0.007 (0.016)
  2 hours postdose (n=79, 79, 79, 79) | 0.136 (0.018) | 0.126 (0.018) | 0.135 (0.018) | 0.019 (0.018)
  4 hours postdose (n=79, 79, 79, 79) | 0.136 (0.018) | 0.115 (0.018) | 0.118 (0.018) | 0.005 (0.018)
  8 hours postdose (n=79, 79, 79, 79) | 0.108 (0.018) | 0.093 (0.018) | 0.087 (0.017) | -0.012 (0.018)
  12 hours postdose (n=78, 79, 78, 79) | 0.092 (0.019) | 0.046 (0.018) | 0.059 (0.018) | -0.033 (0.019)

5. Secondary Outcome: AUC (0-12h) of the Change From Baseline in FEV1 After a Single Dose of MF/F With Spacer Compared to F DPI
Description: as for outcome 1
Time Frame: Up to 12 hours postdose
Population: Participants who received each assigned single-dose treatment, performed at least the 0- and 2-hour spirometry evaluations and met the following criteria: did not use any prohibited concomitant medications; demonstrated satisfactory use of inhaler, space and spirometry maneuvers; and used >80% of prescribed MF DPI across the entire study treatment
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | MF/F MDI With Spacer | F DPI
Number analyzed (Participants) | 79 | 79
Liters | 0.115 (0.016) | 0.097 (0.016)
Statistical Analysis 1: Comparison: MF/F MDI With Spacer vs F DPI; Pairwise Treatment Comparison of MF/F MDI with spacer and F DPI. Analysis was performed using an ANCOVA model extracting the effects due to treatment, sequence, subject (random effect nested within sequence), period, age groups (5 to 7 years and 8 to 11 years) and Baseline FEV1 as a covariate; Test type: Superiority or Other; p = 0.229, ANCOVA; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.012 to 0.048]

6. Secondary Outcome: AUC (0-12h) of the Change From Baseline in FEV1 After a Single Dose of MF/F Without Spacer Compared to F DPI
Description: as for outcome 1
Time Frame: Up to 12 hours postdose
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | MF/F MDI Without Spacer | F DPI
Number analyzed (Participants) | 79 | 79
Liters | 0.093 (0.016) | 0.097 (0.016)
Statistical Analysis 1: Comparison: MF/F MDI Without Spacer vs F DPI; Pairwise Treatment Comparison of MF/F MDI without spacer and F DPI. Analysis was performed using an ANCOVA model extracting the effects due to treatment, sequence, subject (random effect nested within sequence), period, age groups (5 to 7 years and 8 to 11 years) and Baseline FEV1 as a covariate; Test type: Superiority or Other; p = 0.790, ANCOVA; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.033 to 0.025]

7. Secondary Outcome: AUC (0-12h) of the Change From Baseline in FEV1 After a Single Dose of F DPI Compared to Placebo MDI Combined With or Without Spacer
Description: as for outcome 1
Time Frame: Up to 12 hours postdose
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | F DPI | Placebo MDI With or Without Spacer
Number analyzed (Participants) | 79 | 79
Liters | 0.097 (0.016) | -0.009 (0.016)
Statistical Analysis 1: Comparison: F DPI vs Placebo MDI With or Without Spacer; Pairwise Treatment Comparison of F DPI and Placebo MDI combined with or without spacer. Analysis was performed using an ANCOVA model extracting the effects due to treatment, sequence, subject (random effect nested within sequence), period, age groups (5 to 7 years and 8 to 11 years) and Baseline FEV1 as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.106, 95% CI 2-sided [0.077 to 0.135]

8. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) After a Single Dose of MF/F MDI With Spacer, MF/F MDI Without Spacer, F DPI or Placebo MDI Combined With or Without Spacer at 5 and 30 Minutes, 1, 2, 4, 8 and 12 Hours Postdose
Description: Baseline was defined as the average of 2 predose FVC measurements (taken 30 minutes and immediately before dosing).
Time Frame: Baseline and 5 and 30 minutes, 1, 2, 4, 8 and 12 hours postdose
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | MF/F MDI With Spacer | MF/F MDI Without Spacer | F DPI | Placebo MDI With or Without Spacer
Number analyzed (Participants) | 79 | 79 | 79 | 79
Liters
  Baseline (n=79, 79, 79, 79) | 1.914 (0.061) | 1.931 (0.061) | 1.928 (0.061) | 1.913 (0.061)
  5 minutes postdose (n=79, 79, 79, 79) | 0.028 (0.012) | 0.005 (0.012) | 0.032 (0.012) | 0.018 (0.012)
  30 minutes postdose (n=79, 79, 79, 79) | 0.037 (0.013) | 0.020 (0.013) | 0.017 (0.013) | 0.009 (0.013)
  1 hour postdose (n=79, 79, 79, 79) | 0.048 (0.015) | 0.027 (0.014) | 0.022 (0.014) | -0.003 (0.014)
  2 hours postdose (n=79, 79, 79, 79) | 0.023 (0.015) | 0.026 (0.015) | 0.047 (0.015) | 0.015 (0.015)
  4 hours postdose (n=79, 79, 79, 79) | 0.031 (0.015) | 0.018 (0.015) | 0.008 (0.015) | -0.006 (0.015)
  8 hours postdose (n=79, 79, 79, 79) | -0.001 (0.016) | 0.007 (0.015) | -0.013 (0.015) | -0.006 (0.015)
  12 hours postdose (n=78, 79, 78, 79) | -0.001 (0.017) | -0.022 (0.016) | -0.014 (0.016) | -0.012 (0.016)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 30 days after last dose of study drug (up to a total of 90 days)
Description: The Safety Population consisted of all randomized participants who received at least one dose of the study drug.
Arm/Group | MF/F MDI With Spacer | MF/F MDI Without Spacer | F DPI | Placebo MDI With or Without Spacer
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/91 | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/88 | 0/91 | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.